CLINICAL TRIAL: NCT04428333
Title: A Randomized, Double-Blind, Adaptive, Phase II/III Study of GSK3359609 in Combination With Pembrolizumab and 5FU-Platinum Chemotherapy Versus Placebo in Combination With Pembrolizumab Plus 5FU-Platinum Chemotherapy for First-Line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study of GSK3359609 With Pembrolizumab and 5-fluorouracil (5-FU)-Platinum Chemotherapy in Participants With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Acronym: INDUCE-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was stopped by the sponsor based on assessment of the clinical data
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 209227; 2019-003981-42 (EudraCT Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms, Head and Neck
Keywords: GSK3359609; Pembrolizumab; Programmed cell death receptor 1; Inducible T cell co-stimulatory receptor; Keynote-A02; Phase II/III; Platinum-based chemotherapy; 5FU; Head and neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Platinum Compounds; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This will be a randomized, parallel group treatment study with eligible participants receiving either GSK3359609 in combination with pembrolizumab and 5FU-platinum chemotherapy or placebo in combination with pembrolizumab and 5FU-platinum chemotherapy.
Who Masked: Participant, Investigator
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Feladilimab + Pembrolizumab + 5-FU-platinum chemotherapy (Experimental)
  Interventions: Drug: Feladilimab; Drug: Pembrolizumab; Drug: Platinum based chemotherapy; Drug: Fluorouracil (5FU)
- Placebo + Pembrolizumab + 5-FU-platinum chemotherapy (Placebo Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Placebo; Drug: Platinum based chemotherapy; Drug: Fluorouracil (5FU)

INTERVENTIONS:
Drug: Feladilimab — Humanized anti-inducible T cell co-stimulatory receptor (ICOS) immunoglobulin G4 (IgG4) monoclonal antibody (mAb)
  Arms: Feladilimab + Pembrolizumab + 5-FU-platinum chemotherapy
Drug: Pembrolizumab — Humanized anti- programmed cell death receptor1 (anti-PD-1) IgG4 mAb
Drug: Placebo — Sterile normal saline
  Arms: Placebo + Pembrolizumab + 5-FU-platinum chemotherapy
Drug: Platinum based chemotherapy — Cisplatin/carboplatin
Drug: Fluorouracil (5FU) — 5-fluorouracil

SUMMARY:
The purpose of this study is to evaluate if the addition of GSK3359609 to pembrolizumab in combination with 5FU-platinum based chemotherapy improves the efficacy of the pembrolizumab combination with 5FU-platinum based chemotherapy in participants with recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC). This randomized, double-blinded, Phase II/III study will compare the combination of GSK3359609 with pembrolizumab and 5FU-platinum chemotherapy to placebo in combination with pembrolizumab and 5FU-platinum chemotherapy in participants with recurrent or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx or larynx.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Male or female, age >=18 years
* HNSCC that was diagnosed as recurrent or metastatic and considered incurable by local therapies.
* Primary tumor location of the oral cavity, oropharynx, hypopharynx or larynx.
* No prior systemic therapy administered in the recurrent or metastatic setting (with the exception of systemic therapy completed >6 months prior if given as part of multimodal treatment for locally advanced disease and no disease progression/recurrence within 6 months of the completion of curatively intended systemic treatment).
* Measurable disease per RECIST version 1.1 guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* Adequate organ function.
* Life expectancy of at least 12 weeks.
* Female participants: must not be pregnant, not breastfeeding, and be either not a woman of childbearing potential (WOCBP); or be a WOCBP who agrees to use a highly effective method of birth control from 30 days prior to randomization and for at least 120 days after the last dose of study treatment.
* Male participants with female partners of child-bearing potential: must agree to use a highly effective contraception while receiving study treatment and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this periods.
* Provide tumor tissue from excisional or core biopsy (fine needle aspirates and bone biopsies are not acceptable) acquired within 2 years prior to randomization for PD-L1 immunohistochemistry (IHC) testing by central laboratory.
* Have PD-L1 IHC CPS status by central laboratory testing.
* Have results from testing of human papilloma virus (HPV) status for oropharyngeal cancer.

Exclusion Criteria:

* Prior therapy with an anti-PD-1/L1/L2, anti-Inducible T Cell Co-Stimulatory Receptor (ICOS) directed agent.
* Systemic approved or investigational anticancer therapy within 30 days or 5 half lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the date of randomization. - Has high risk of bleeding (examples include but not limited to tumors encasing or infiltrating a major vessel [i.e. carotid, jugular, bronchial artery] and/or exhibits other high-risk features such as an arteriovenous fistula)
* Active tumor bleeding - Grade 3 or Grade 4 hypercalcemia.
* Major surgery less than or equal to (<=) 28 days prior to randomization.
* Participants must have also fully recovered from any surgery (major or minor) and/or its complications before randomization
* Toxicity from previous anticancer treatment that includes: a. Grade 3/Grade 4 toxicity considered related to prior immunotherapy and that led to treatment discontinuation and b. toxicity related to prior treatment that has not resolved to <=Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <=Grade 2).
* Received transfusion of blood products or administration of colony stimulating factors within 14 days prior to randomization.
* Central nervous system (CNS) metastases, with the following exception: Participants with asymptomatic CNS metastases who are clinically stable and have no requirement for steroids for at least 14 days prior to randomization.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last 3 years with the exception of: a. any other invasive malignancy for which the participant was definitively treated, has been disease-free for <=3 years. b. curatively treated non-melanoma skin cancer or successfully treated in situ carcinoma and/or. c. low-risk early stage prostate cancer defined as: Stage T1c or T2a with a Gleason score <=6 and prostatic-specific antigen less than (<)10 nanograms per milliliter (ng/mL) either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to randomization.
* Autoimmune disease or syndrome that required systemic treatment within the past 2 years.
* Has a diagnosis of immunodeficiency or is receiving systemic steroids (>10 milligram [mg] oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to randomization.
* Receipt of any live vaccine within 30 days prior randomization.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* Has current pneumonitis or history of non-infectious pneumonitis that required steroids or other immunosuppressive agents.
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions.
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* Recent history of allergen desensitization therapy within 4 weeks of randomization.
* History or evidence of cardiac abnormalities within the 6 months prior to randomization which include: a. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third-degree atrioventricular block. b. Cardiomyopathy, myocardial infarction, acute coronary syndromes(including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting. c. Congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system. d. Symptomatic pericarditis.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy.
* Known human immunodeficiency virus (HIV) infection, or positive test for hepatitis B active infection (presence of hepatitis B surface antigen), or hepatitis C active infection.
* History of severe hypersensitivity to monoclonal antibodies or to the chemotherapies under investigation including any ingredient used in the formulation.
* Known history of active tuberculosis.
* Any serious (>=Grade 3) and/or unstable pre-existing medical condition (aside from malignancy).
* Any psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the date of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- GSK Investigational Site, Duarte, California, United States
- Argentina (4):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Oro Verde Entre RIos
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (4):
  - GSK Investigational Site, Blacktown
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Melbourne
  - GSK Investigational Site, Woolangabba
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
- Brazil (3):
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Copenhagen, Denmark
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Strasbourg
- Germany (4):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Ulm
- GSK Investigational Site, Dublin, Ireland
- Italy (6):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Savona
- Japan (2):
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Tomaszów Mazowiecki
  - GSK Investigational Site, Warsaw
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Suceava
- GSK Investigational Site, Pushkin, Russia
- South Korea (5):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Stockholm, Sweden
- United Kingdom (3):
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in the study stopped following the review of unblinded interim safety and efficacy data by IDMC, after a pre-specified futility analysis of the 209229(NCT04128696) trial. A Dear investigator letter (DIL) was issued to stop screening & randomization of more participants in both studies. Participants discontinued feladilimab/placebo, but treatment with pembrolizumab plus fluorouracil (5FU) platinum chemotherapy continued until disease progression, death or unacceptable toxicity.
Pre-assignment Details: One participant was incorrectly re-randomized into the study twice and was given a new participant ID. However, the participant was considered only once for the analyses. An additional participant was randomized after the data cut off for the primary posting and received only pembrolizumab. Therefore, this participant is included in safety analysis for the end of study posting.
Groups:
- Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy: Participants were administered feladilimab (humanized anti- ICOS IgG4 mAb) and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an IV infusion along with 5 FU-platinum chemotherapy (cisplatin OR carboplatin) Q3W.
- Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy: Participants were administered placebo and pembrolizumab as an IV infusion along with 5 FU-platinum chemotherapy (cisplatin OR carboplatin) Q3W.
Period: Overall Study
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Started | 57 | 60
Modified Intent-to-Treat (mITT) Population (5 participants initially randomized to feladilimab + chemotherapy arm and 5 participants initially randomized to placebo + chemotherapy arm were dosed only after DIL date requesting immediate discontinuation of feladilimab/placebo and were not included in the mITT population.) | 52 | 55
Safety Population (6 participants were initially randomized to feladilimab+pembrolizumab+5-FU-platinum chemotherapy arm but never received feladilimab. 5 of them were dosed after the DIL date and reassigned to the placebo+pembrolizumab+5-FU-platinum chemotherapy arm. 1 participant was initially randomized to feladilimab+pembrolizumab+5-FU-platinum chemotherapy arm but never dosed. An additional participant,randomized post-data cut off,received only pembrolizumab and is included in the end of study safety analysis.) | 51 | 65
Completed | 37 | 35
Not Completed | 20 | 25
Not completed — Physician Decision | 5 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Study Terminated By Sponsor | 14 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 37 | 40 | 77
  >=65-84 years | 20 | 20 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 47 | 46 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 2 | 1 | 3
  Asian - East Asian Heritage | 5 | 7 | 12
  Asian - Japanese Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 2 | 1 | 3
  Black or African American | 1 | 0 | 1
  Missing | 2 | 1 | 3
  White - White/Caucasian/European Heritage | 43 | 50 | 93

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in mITT Population
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Kaplan-Meier estimate for the median OS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: mITT population: All randomized participants whether or not randomized intervention was administered, excluding those who were first dosed or randomized after the date of DIL requesting immediate discontinuation of feladilimab /placebo. Participants were analyzed based on the study intervention to which the participant was randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Months | NA [5.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [4.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The hazard ratio and corresponding 2-sided 95% confidence interval was calculated from the cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20 vs. CPS <1) and Human Papilloma Virus (HPV) status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Superiority — Other; p = 0.740, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the one sided log-rank test, stratified by stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20 vs. CPS <1) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 2.16, 95% CI 2-sided [0.20 to 23.87]

2. Primary Outcome: OS in Programmed Death Receptor-ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1 Population
Description: OS was defined as the time from the date of randomization until the date of death due to any cause. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median OS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Months | NA [5.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [4.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The hazard ratio and corresponding 2-sided 95% confidence interval was calculated from the cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by PD-L1 expression (CPS ≥ 20 vs 1≤ CPS<20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Superiority — Other; p = 0.740, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the one sided log-rank test, stratified by stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 2.16, 95% CI 2-sided [0.20 to 23.87]

3. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1 in mITT Population
Description: PFS per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 was defined as the time from the date of randomization to the date of first documented disease progression or death due to any cause, whichever occurs first. Kaplan-Meier estimate for the median PFS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: All participants in the mITT population were analyzed
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Months | 5.5 [3.7 to 5.5] | 4.7 [4.7 to 5.6]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The hazard ratio and corresponding 2-sided 95% confidence interval was calculated from the cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20 vs. CPS <1) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Superiority — Other; p = 0.284, Stratified Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.20 to 2.43]

4. Secondary Outcome: PFS Per RECIST v1.1 in the PD-L1 CPS ≥1 Population
Description: PFS per RECIST v1.1 was defined as the time from the date of randomization until the date of disease progression or death due to any cause, whichever occurs first. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median PFS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Months | 5.5 [3.7 to 5.5] | 4.7 [4.7 to 6.1]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The hazard ratio and corresponding 2-sided 95% confidence interval was calculated from the cox regression model with Efron's method of tie handling with treatment as a covariate and stratified by PD-L1 expression (CPS≥20 vs 1≤CPS<20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Superiority — Other; p = 0.284, Stratified Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.20 to 2.43]

5. Secondary Outcome: Milestone OS Rate at 12, 24 and 36 Months in mITT Population
Description: Milestone OS rate at 12, 24, and 36 months was not evaluated.
Time Frame: Months 12, 24 and 36
Population: mITT population. All participants were on study for <12 months. The maximum duration of follow-up was approximately 7 months.
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Milestone OS Rate at 12, 24 and 36 Months in PD-L1 CPS ≥1 Population
Description: Milestone OS rate at 12, 24, and 36 months was not evaluated. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Months 12, 24 and 36
Population: Data for participants with PD-L1 CPS ≥1 in mITT population were to be presented. All participants were on study for <12 months. The maximum duration of follow-up was approximately 7 months.
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR) Per RECIST v1.1 in mITT Population
Description: ORR per RECIST v1.1 was defined as the proportion of the participants who have a complete response (CR) or partial response (PR) as the best overall response per RECIST v1.1 based upon investigator assessment. As a randomized double-blind study in which primary endpoints are OS and PFS, the confirmation of CR and PR was not required. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted.
Time Frame: Up to approximately 7 months
Population: All participants in the mITT population were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Percentage of participants | 19.2 [9.6 to 32.5] | 23.6 [13.2 to 37.0]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The comparison between treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20 vs. CPS <1) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -4.8, 95% CI 2-sided [-20.8 to 11.3]

8. Secondary Outcome: ORR Per RECIST v1.1 in PD-L1 CPS ≥1 Population
Description: ORR per RECIST v1.1 was defined as the proportion of the participants who have a complete response (CR) or partial response (PR) as the best overall response per RECIST v1.1 based upon investigator assessment. As a randomized double-blind study in which primary endpoints are OS and PFS, the confirmation of CR and PR was not required. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in mITT population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Percentage of participants | 18.4 [8.8 to 32.0] | 23.1 [12.5 to 36.8]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The comparison between treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included PD-L1 expression (CPS≥20 vs 1≤CPS<20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -5.1, 95% CI 2-sided [-21.4 to 11.3]

9. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 in mITT Population
Description: DCR per RECIST v1.1 based upon investigator assessment, was defined as the percentage of participants with a best overall response of CR or PR at any time plus stable disease (SD) meeting the minimum time of 15 weeks. A status of SD≥15 weeks will be assigned if the follow-up disease assessment has met the SD criteria at least once after the date of randomization at a minimum of 14 weeks (98 days) considering a one-week visit window. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted.
Time Frame: Up to approximately 7 months
Population: All participants in the mITT population were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Percentage of participants | 32.7 [20.3 to 47.1] | 36.4 [23.8 to 50.4]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Other; Difference in Percentage = -4.8, 95% CI 2-sided [-22.2 to 13.1]

10. Secondary Outcome: DCR Per RECIST v1.1 in PD-L1 CPS ≥1 Population
Description: DCR per RECIST v1.1 based upon investigator assessment, was defined as the percentage of participants with a best overall response of CR or PR at any time plus stable disease (SD) meeting the minimum time of 15 weeks. A status of SD≥15 weeks will be assigned if the follow-up disease assessment has met the SD criteria at least once after the date of randomization at a minimum of 14 weeks (98 days) considering a one-week visit window. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in mITT population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Percentage of participants | 30.6 [18.3 to 45.4] | 34.6 [22.0 to 49.1]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; The comparison between treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -5.1, 95% CI 2-sided [-22.8 to 13.3]

11. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1 in mITT Population
Description: DoR per RECIST v1.1 is defined as the time from first documented evidence of CR or PR until first documented disease progression per RECIST v1.1 based upon investigator assessment or death due to any cause, whichever occurs first, among participants who demonstrated CR or PR as the best overall response per RECIST v1.1. Kaplan-Meier estimate for the median DoR is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: Data for participants with a best overall response of CR or PR in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 10 | 13
Months | NA [NA to NA] — The median was not reached at the time of primary completion date. The upper and lower limit of the 95% CI was not calculable from the available data at the time of data cut off. | 2.8 [1.2 to 2.8]

12. Secondary Outcome: DoR Per RECIST v1.1 in PD-L1 CPS ≥1 Population
Description: DoR per RECIST v1.1 is defined as the time from first documented evidence of CR or PR until first documented disease progression per RECIST v1.1 based upon investigator assessment or death due to any cause, whichever occurs first, among participants who demonstrated CR or PR as the best overall response per RECIST v1.1. Kaplan-Meier estimate for the median DoR is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 7 months
Population: Data for participants with a best overall response of CR or PR in mITT population with PD-L1 CPS ≥1 are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 9 | 12
Months | NA [NA to NA] — The median was not reached at the time of primary completion date. The upper and lower limit of the 95% CI was not calculable from the available data at the time of data cut off. | 2.8 [1.4 to 2.8]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) in Safety Population
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention
Time Frame: Up to approximately 37.2 months
Population: Safety Population: All randomized participants who took at least 1 dose of study intervention. Participants were analyzed according to the actual study intervention received. An additional participant was randomized after the data cut off and received pembrolizumab. Therefore, participant was included in safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants | 51 | 65

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Safety Population
Description: SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and other situations according to medical or scientific judgement.
Time Frame: Up to approximately 37.2 months
Population: Safety Population. An additional participant was randomized after the data cut-off and received pembrolizumab. Therefore, this participant was included in safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants | 23 | 32

15. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) in Safety Population
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs).
Time Frame: Up to approximately 37.2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants | 29 | 43

16. Secondary Outcome: Number of Participants With AEs in Programmed Death Ligand-1 (PD-L1) Combined Positive Score (CPS ≥1) Population
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 37.2 months
Population: Data for participants with PD-L1 CPS ≥1 in the safety population are presented. An additional participant was randomized after the data cut-off and received pembrolizumab. Therefore, this participant was included in safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 48 | 62

17. Secondary Outcome: Number of Participants With SAEs in PD-L1 CPS ≥1 Population
Description: SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and other situations according to medical or scientific judgement. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 21 | 32

18. Secondary Outcome: Number of Participants With AESIs in PD-L1 CPS ≥1 Population
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 27 | 40

19. Secondary Outcome: Severity of AEs in Safety Population
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity for each AE was reported during the study and assigned a grade according to the NCI-CTCAE v5.0. from Grade 1 through Grade 5. Grade 1= mild toxicity; Grade 2 = moderate toxicity; Grade 3 = severe toxicity; Grade 4 = life-threatening or disabling toxicity, Grade 5 = death related to toxicity.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants
  Grade 1 | 1 | 3
  Grade 2 | 17 | 15
  Grade 3 | 23 | 34
  Grade 4 | 4 | 10
  Grade 5 | 6 | 3

20. Secondary Outcome: Severity of SAEs in Safety Population
Description: A SAE was defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement. Severity for each SAE was reported during the study and assigned a grade according to the NCI-CTCAE v5.0. from Grade 1 through Grade 5. Grade 1= mild toxicity; Grade 2 = moderate toxicity; Grade 3 = severe toxicity; Grade 4 = life-threatening or disabling toxicity, Grade 5 = death related to toxicity. Data of participants experiencing SAEs of Grade >= 3 has been presented.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants | 17 | 26

21. Secondary Outcome: Severity of AESIs in Safety Population
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). Severity of each AESI was reported during the study and was assigned a grade according to the NCI-CTCAE. AESIs severity were graded on a 5-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, 3 = severe; inability to work or perform normal daily activity, 4 = life-threatening consequences and 5 = death related to AE. Data of participants experiencing AESIs of Grade >= 3 have been presented.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 51 | 65
Participants | 5 | 4

22. Secondary Outcome: Severity of AEs in PD-L1 CPS ≥1 Population
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity for each AE was reported during the study and assigned a grade according to the NCI-CTCAE v5.0. from Grade 1 through Grade 5. Grade 1= mild toxicity; Grade 2 = moderate toxicity; Grade 3 = severe toxicity; Grade 4 = life-threatening or disabling toxicity, Grade 5 = death related to toxicity. Data of participants experiencing AEs of Grade >= 3 have been presented. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 30 | 45

23. Secondary Outcome: Severity of SAEs in PD-L1 CPS ≥1 Population
Description: A SAE was defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement. Severity for each SAE was reported during the study and assigned a grade according to the NCI-CTCAE v5.0. from Grade 1 through Grade 5. Grade 1= mild toxicity; Grade 2 = moderate toxicity; Grade 3 = severe toxicity; Grade 4 = life-threatening or disabling toxicity, Grade 5 = death related to toxicity. Data of participants that experienced SAEs of Grade >= 3 have been presented. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 15 | 26

24. Secondary Outcome: Severity of AESI in PD-L1 CPS ≥1 Population
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). Severity of each AESI was reported during the study and was assigned a grade according to the NCI-CTCAE. AESIs severity were graded on a 5-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, 3 = severe; inability to work or perform normal daily activity, 4 = life-threatening consequences and 5 = death related to AE. Data of participants that experienced AESIs of Grade >= 3 have been presented.
Time Frame: Up to approximately 37.2 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 48 | 62
Participants | 5 | 4

25. Secondary Outcome: Number of Participants With Dose Modifications in Safety Population
Description: Number of participants with dose modifications (including dose interruptions, dose delays, dose reductions and treatment discontinuations) were reported by each interventional component.
Time Frame: Up to approximately 7 months
Population: All participants in the safety population were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 50 | 65
Participants
  Dose interruption per component - feladilimab | 0 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose interruption per component - placebo | NA — Participants in this treatment arm were not dosed with placebo | 0
  Dose interruption per component - pembrolizumab | 0 | 0
  Dose interruption per component - carboplatin/cisplatin | 1 | 1
  Dose interruption per component - fuorouracil | 0 | 7
  Dose delays per component - feladilimab | 13 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose delays per component - placebo | NA — Participants in this treatment arm were not dosed with placebo | 12
  Dose delays per component - pembrolizumab | 13 | 13
  Dose delays per component - cisplatin/carboplatin | 12 | 9
  Dose delays per component - fluorouracil | 9 | 10
  Dose Reduction per component - feladilimab | NA — Dose reductions were not permitted for feladilimab | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose Reduction per component - placebo | NA — Participants in this treatment arm were not dosed with placebo | NA — Dose reductions were not permitted for placebo
  Dose Reduction per component - pembrolizumab | NA — Dose reductions were not permitted for pembrolizumab | NA — Dose reductions were not permitted for pembrolizumab
  Dose Reduction per component - carboplatin/cisplatin | 12 | 19
  Dose Reduction per component - fluorouracil | 18 | 21
  Treatment discontinuation per component - feladilimab/placebo | 50 | 56
  Treatment discontinuation per component - pembrolizumab | 10 | 15
  Treatment discontinuation per component - carboplatin/cisplatin | 16 | 18
  Treatment discontinuation per component - fluorouracil | 13 | 18

26. Secondary Outcome: Number of Participants With Dose Modifications in PD-L1 CPS ≥1 Population
Description: Number of participants with dose modifications (including dose interruptions, dose delays, dose reductions and treatment discontinuations) were reported by each interventional component. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in the safety population are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 47 | 62
Participants
  Dose Interruptions per component- feladilimab | 0 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose Interruptions per component- placebo | NA — Participants in this treatment arm were not dosed with placebo | 0
  Dose Interruptions per component- pembrolizumab | 0 | 0
  Dose Interruptions per component- carboplatin/cisplatin | 1 | 1
  Dose Interruptions per component- fluorouracil | 0 | 7
  Dose Delays per component - feladilimab | 12 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose Delays per component - placebo | NA — Participants in this treatment arm were not dosed with placebo | 11
  Dose Delays per component - pembrolizumab | 2 | 12
  Dose Delays per component - carboplatin/cisplatin | 11 | 9
  Dose Delays per component - fluorouracil | 8 | 9
  Dose Reductions per component - feladilimab | NA — Dose reductions were not permitted for feladilimab | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose Reductions per component - placebo | NA — Participants in this treatment arm were not dosed with placebo | NA — Dose reductions were not permitted for placebo
  Dose Reductions per component - pembrolizumab | NA — Dose reductions were not permitted for pembrolizumab | NA — Dose reductions were not permitted for pembrolizumab
  Dose Reductions per component - carboplatin/cisplatin | 11 | 16
  Dose Reductions per component - fluorouracil | 16 | 19
  Treatment Discontinuations per component - feladilimab/placebo | 47 | 53
  Treatment Discontinuations per component - pembrolizumab | 10 | 14
  Treatment Discontinuations per component - carboplatin/cisplatin | 13 | 16
  Treatment Discontinuations per component - fluorouracil | 15 | 16

27. Secondary Outcome: Time to Deterioration (TTD) in Pain in mITT Population
Description: TTD in pain is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the European Organization for Research and Treatment of Cancer Item Library(EORTC IL51) Questionnaire pain domain, i.e. an increase from baseline of at least 8.33 observed at all subsequent non-missing visits. The EORTC Quality of Life Questionnaire 35-Item Head and Neck Module (QLQ-H&N35) is a head and neck specific module with multi-item scales. The mouth pain, swallowing, speech problems, opening mouth, coughing, feeding tube, and trouble with social eating domains were administered and referred to as the EORTC IL51. The questionnaire scores for each scale and single-item measure are averaged and transformed linearly to present a score ranging from 0-100. A high score represents a high/healthy level of functioning. Kaplan-Meier estimate for the median TTD is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 7 months
Population: All participants in the mITT population were analyzed
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Months | 4.4 [2.1 to 4.4] | 2.8 [1.4 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Other; p = 0.329, Stratified Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.42 to 1.71]

28. Secondary Outcome: TTD in Pain in PD-L1 CPS ≥1 Population
Description: TTD in pain is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the EORTC IL51 pain domain, i.e. an increase from baseline of at least 8.33 observed at all subsequent non-missing visits. The EORTC QLQ-H&N35 is a head and neck specific module with multi-item scales. The mouth pain, swallowing, speech problems, opening mouth, coughing, feeding tube, and trouble with social eating domains were administered and referred to as the EORTC IL51. The questionnaire scores for each scale and single-item measure are averaged and transformed linearly to present a score ranging from 0-100. A high score represents a high/healthy level of functioning. Kaplan-Meier estimate for the median TTD is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells to the total number of viable tumor cells.
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in the mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Months | 3.4 [1.3 to 4.4] | 2.8 [1.4 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — Other; p = 0.302, Stratified Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.40 to 1.69]

29. Secondary Outcome: TTD in Physical Function in mITT Population
Description: TTD in physical function (PF) is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the PF T-score, i.e. a decrease from baseline of at least 2.4 observed at all subsequent non-missing visits, as measured by the Patient-Reported Outcomes Measurement Information System - Physical Function (PROMIS PF 8c).The PROMIS PF 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It includes a 5-point scale with three sets of response options. Scores on the PROMIS PF 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning.
Time Frame: Up to approximately 7 months
Population: All participants in the mITT population were analyzed
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 52 | 55
Months | 2.8 [1.4 to NA] — The available data does not allow for the calculation of the upper limit of the 95% CI. | 4.3 [2.1 to 5.6]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Other; p = 0.472, Stratified Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.44 to 2.11]

30. Secondary Outcome: TTD in Physical Function in PD-L1 CPS ≥1 Population
Description: TTD in PF is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the PF T-score, i.e. a decrease from baseline of at least 2.4 observed at all subsequent non-missing visits, as measured by the PROMIS PF 8c.The PROMIS PF 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It includes a 5-point scale with three sets of response options. Scores on the PROMIS PF 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells
Time Frame: Up to approximately 7 months
Population: Data for participants with PD-L1 CPS ≥1 in the mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
Number analyzed (Participants) | 49 | 52
Months | 4.8 [2.1 to NA] — The available data does not allow for the calculation of the upper limit of the 95% CI. | 4.3 [2.1 to 5.6]
Statistical Analysis 1: Comparison: Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy vs Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — Other; p = 0.335, Stratified Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.36 to 1.90]

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected from Day 1 to up to approximately 37.2 months.
Description: 6 participants were initially randomized to feladilimab+pembrolizumab+5-FU-platinum chemotherapy arm but never received feladilimab. 5 of them were dosed after the DIL date and reassigned to the placebo+pembrolizumab+5-FU-platinum chemotherapy arm. 1 participant was initially randomized to feladilimab+pembrolizumab+5-FU-platinum chemotherapy arm but never dosed. An additional participant,randomized post-data cut off,received only pembrolizumab and is included in the end of study safety analysis.
Arm/Group | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy
All-Cause Mortality (participants affected / at risk) | 33/51 | 39/65
Serious Adverse Events (participants affected / at risk) | 23/51 | 32/65
Other Adverse Events (participants affected / at risk) | 50/51 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy (N=51) | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 1 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheostomy infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Embedded device (Product Issues) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feladilimab + Pembrolizumab + 5-FU-platinum Chemotherapy (N=51) | Placebo + Pembrolizumab + 5-FU-platinum Chemotherapy (N=65)
Anaemia (Blood and lymphatic system disorders) | 27 (40) | 30 (53)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 7 (14)
Neutropenia (Blood and lymphatic system disorders) | 9 (15) | 21 (47)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8) | 17 (29)
Constipation (Gastrointestinal disorders) | 13 (15) | 16 (16)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 21 (37)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 8 (9)
Nausea (Gastrointestinal disorders) | 22 (27) | 32 (40)
Stomatitis (Gastrointestinal disorders) | 12 (12) | 16 (21)
Vomiting (Gastrointestinal disorders) | 8 (9) | 13 (23)
Asthenia (General disorders) | 8 (12) | 13 (15)
Fatigue (General disorders) | 17 (20) | 24 (29)
Mucosal inflammation (General disorders) | 6 (6) | 16 (20)
Pyrexia (General disorders) | 4 (6) | 7 (11)
Oral candidiasis (Infections and infestations) | 2 (2) | 9 (11)
Blood creatinine increased (Investigations) | 3 (3) | 10 (21)
Neutrophil count decreased (Investigations) | 10 (18) | 10 (16)
Platelet count decreased (Investigations) | 6 (8) | 9 (11)
Weight decreased (Investigations) | 8 (8) | 5 (5)
White blood cell count decreased (Investigations) | 5 (13) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 7 (7)
Headache (Nervous system disorders) | 5 (5) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (5)
Oral pain (Gastrointestinal disorders) | 3 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 3 (3) | 3 (3)
Lymphocyte count decreased (Investigations) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (7)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 4 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 6 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
COVID-19 (Infections and infestations) | 2 (2) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6)
Pneumonia (Infections and infestations) | 1 (1) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Hypothyroidism (Endocrine disorders) | 7 (10) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8)
Hypertension (Vascular disorders) | 3 (4) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT04428333/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04428333/SAP_001.pdf